CLINICAL TRIAL: NCT02367521
Title: Repetitive Transcranial Magnetic Stimulation (rTMS) for the Treatment of Depression & Other Neuropsychiatric Symptoms After Traumatic Brain Injury (TBI)
Acronym: rTMS TBI
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NA_00090926
Record Dates: First submitted 2015-02-09; First posted 2015-02-20 (Estimated); Results first posted 2018-08-31 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: TBI Depression
Keywords: TBI Depression; co-morbid psychiatric symptoms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- LFR rTMS (Experimental): Investigators propose to deliver 1200 pulses daily at 110% Motor threshold for 4 weeks using four trains of 300 pulses daily separated by an intertrain interval of 60 seconds.
  Interventions: Combination Product: Low Frequency Right sided repetitive transcranial magnetic stimulation (LFR rTMS)
- Sham Treatment (Placebo Comparator): Control patients will receive treatment using an identically appearing coil that produces the same sound and is the same weight as the active coil, but has negligible magnetic field strength
  Interventions: Device: Sham Comparator: Sham Treatment

INTERVENTIONS:
Combination Product: Low Frequency Right sided repetitive transcranial magnetic stimulation (LFR rTMS) — LFR rTMS will be delivered at the Brain Stimulation Program at The Johns Hopkins Hospital with a Magstim Super Rapid 2 stimulator with a focal double 70-mm air cooled coil. LFR rTMS will be administered to the Experimental Group.
  Control patients will receive treatment using an identically appearing coil that produces the same sound and is the same weight as the active coil, but has negligible magnetic field strength.
  Other Names: low frequency right rTMS
  Arms: LFR rTMS
Device: Sham Comparator: Sham Treatment — Control patients will receive treatment using an identically appearing coil that produces the same sound and is the same weight as the active coil, but has negligible magnetic field strength
  Other Names: Placebo
  Arms: Sham Treatment

SUMMARY:
Traumatic brain injury (TBI) is frequently complicated by depression and other problems such as post traumatic stress disorder (PTSD), sleep disturbance, cognitive deficits and behavioral problems. Untreated depression can lead to reduced productivity and poor global outcome. There is no Food and Drug Administration (FDA) approved drug for the treatment of TBI-related depression. The overarching goal of this small study is to determine the effectiveness of low frequency right (LFR) rTMS for the treatment of post-TBI depression and co-occurring psychiatric symptoms. Repetitive transcranial magnetic stimulation (rTMS) is a brain stimulation technique. It involves generating a brief magnetic field in a coil that is placed on the scalp. The magnetic field passes through the skull and induces a weak electrical current in the brain that briefly activates neural circuits at the stimulation site. Adults aged 18 and older, with a history of head injury of mild or moderate severity , who are currently experiencing symptoms of clinical depression may join the study.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 and over
2. H/o closed head injury
3. Must meet Department of Defense (DoD) criteria for mild or moderate Traumatic Brain Injury (TBI)
4. Must meet criteria for major depression as assessed by the Structured Clinical Interview (SCID) for Diagnostic and Statistical Manual IV (DSM-IV) and a score greater than 10 on the Hamilton Depression 17 (HAM-D17) Scale

Exclusion Criteria:

1. Subjects with skull fracture
2. Subjects who meet DoD criteria for severe TBI
3. Subjects who are on psychotropics or mood stabilizing medications (e.g. antidepressants, antipsychotics, anxiolytics, sedative/hypnotics.
4. Subjects who are medically unstable
5. History of active substance abuse x 1 month
6. Current psychotic illness
7. Evidence of frontal lesions on brain scan.
8. Individuals with a significant neurological disorders that could increase risk of seizures such as brain tumor, cerebral aneurysm, any h/o seizures and/or family h/o seizures
9. Dementia
10. Mini Mental State Exam score of less than or equal to 24
11. A positive and unmitigated response to any question on the Transcranial Magnetic Stimulation Safety Screen questionnaire
12. Electroconvulsive therapy (ECT) treatment within 6 months prior to the screening visit
13. History of treatment with rTMS therapy for any disorder
14. History of treatment with Vagus Nerve Stimulation (VNS)
15. History of treatment with Deep Brain Stimulation (DBS)
16. Cardiac pacemakers, implanted medication pumps, intracardiac lines,
17. Intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed.
18. Implanted neurostimulators
19. Known or suspected pregnancy
20. Investigators, personnel affiliated with this study, and their immediate families.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-10-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 70 participants passed screening & were enrolled in study. 36 were not randomized.14 lost to follow-up, 5 refused due to scheduling, 5 did not meet DSM IV criteria: major depression, 3 concerns about receiving rTMS, 2 psychotropics, 2 did not have TBI, 1 using illicit drugs, 1 skull fracture, 1 severe TBI, 1 with seizure history, 1 MRI focal lesion
Groups:
- LFR rTMS: Investigators propose to deliver 1200 pulses daily at 110% Motor threshold for 4 weeks using four trains of 300 pulses daily separated by an intertrain interval of 60 seconds.
  Low Frequency Right sided repetitive transcranial magnetic stimulation (LFR rTMS): LFR rTMS will be delivered at the Brain Stimulation Program at The Johns Hopkins Hospital with a Magstim Super Rapid 2 stimulator with a focal double 70-mm air cooled coil. LFR rTMS will be administered to the Experimental Group.
  Control patients will receive treatment using an identically appearing coil that produces the same sound and is the same weight as the active coil, but has negligible magnetic field strength.
Period: Overall Study
Arm/Group | LFR rTMS | Sham Treatment
Started | 17 | 17
Completed | 13 | 17
Not Completed | 4 | 0
Not completed — severe headache after intervention | 2 | 0
Not completed — unable to find transportation | 2 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were only documented and analyzed for participants who complete the study. Details for the four who dropped out are no longer available.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham Treatment | LFR rTMS | Total
Number analyzed (Participants) | 17 | 13 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.2 (14.6) | 39.8 (14.2) | 40 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 11 | 5 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 10 | 9 | 19
  Non-White | 7 | 4 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 13 | 30
Months Depressed Since Injury [Mean (Standard Deviation); unit: months] | 39.4 (43) | 39.6 (36.1) | 39.47 (39.51)

OUTCOME MEASURES:

1. Primary Outcome: Average Depression Score Using the Hamilton Depression (HAM-D) 17 Scale
Description: The HAM-D was used to determine the effectiveness of LFR rTMS for the treatment of post-TBI depression. The scale ranges from 0-54, with 0-7 = Normal; 8-13= Mild Depression; 14-18= Moderate Depression, 19-22= Severe Depression, >/= 23 = Very Severe Depression.
Time Frame: Mean at baseline, 4 weeks, 8 weeks, 12 weeks, and 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LFR rTMS | Sham Treatment
Number analyzed (Participants) | 13 | 17
units on a scale
  Baseline | 23.154 (4.375) | 23.076 (4.356)
  4 weeks | 13.154 (8.444) | 12.706 (6.697)
  8 weeks | 12.538 (9.744) | 12.647 (6.901)
  12 weeks | 14.077 (10.21) | 12.824 (8.435)
  16 weeks | 11.154 (9.529) | 12.941 (8.877)

2. Primary Outcome: Mean Clinical Global Improvement- Severity/Improvement Scale Score (CGI-I/CGI-S)
Description: The CGI scale is broken down into the CGI-S and CGI-I components. CGI-S is the baseline severity of mental illness. 1= normal, not at all ill; 2= borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill patients. The CGI-S is only performed at baseline.
  The CGI-I component (which is any measure after intervention) is as follows: 1=very much improved since the initiation of treatment; 2=much improved; 3=minimally improved; 4=no change from baseline (the initiation of treatment); 5=minimally worse; 6= much worse; 7=very much worse since the initiation of treatment.
Time Frame: Mean at baseline, 4, 8, 12, and 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LFR rTMS | Sham Treatment
Number analyzed (Participants) | 13 | 17
units on a scale
  CGI Baseline (severity) | 4.846 (0.801) | 5 (0.791)
  CGI 4 weeks (improvement) | 2.308 (1.109) | 2.824 (1.334)
  CGI 8 weeks (improvement) | 2.385 (1.044) | 2.471 (1.125)
  CGI 12 weeks (improvement) | 2.385 (1.0444) | 2.588 (1.064)
  CGI 16 weeks (improvement) | 2.077 (0.854) | 2.471 (1.281)

3. Primary Outcome: Mean Suicidal Ideation as Assessed by the Beck Suicidal Ideation Scale (BSSI)
Description: The BSSI scale is used to assess the degree of suicidal ideation. The scale ranges from 0-38, with 0= no suicidality, and 38 = highest severity of suicidal ideation
Time Frame: Mean at baseline, 4, 8, 12, and 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LFR rTMS | Sham Treatment
Number analyzed (Participants) | 13 | 17
units on a scale
  Baseline | 0.462 (1.127) | 1.294 (1.896)
  4 weeks | 0.077 (0.277) | 0.706 (1.359)
  8 weeks | 0.154 (0.376) | 0.353 (0.862)
  12 weeks | 0 (0) | 0.529 (1.007)
  16 weeks | 0.00 (0) | 0.471 (0.943)

4. Secondary Outcome: Ability to Inhibit Cognitive Interference as Assessed by the Stroop Color Word Test (SCWT)
Description: The SCWT is used to assess the ability to inhibit cognitive interference that occurs when the processing of a specific stimulus feature impedes the simultaneous processing of a second stimulus attribute. Participants are required to read three different tables as fast as possible. Two of the tables represent the "congruous condition" in which participants are required to read names of colors printed in black ink and name different color patches. In the third table, "incongruous condition" the color-words are printed in a different color in (ie: the word "red" is printed in green ink). Within this third table, participants are required to name the color of the ink instead of reading the word. The score is based on the number of items completed, which ranges from 0 to 100, with a higher score reflecting a better outcome.
Time Frame: Mean at baseline and 16 weeks
Measure: Mean (Standard Deviation); unit: items completed
Arm/Group | LFR rTMS | Sham Treatment
Number analyzed (Participants) | 13 | 17
items completed
  0 weeks | 43.2 (13.3) | 42.4 (8.2)
  16 weeks | 45.4 (11.9) | 43.1 (11.6)

5. Secondary Outcome: Cognitive Reasoning as Assessed by the Number of Completed Categories on the Wisconsin Card Scoring Test (WCST)
Description: The participant points to choice on the screen and the tester manipulates the mouse to make the response. The participant tells the tester if he or she wants to change the response and the tester clicks on the screen. The score is the number of completed categories, ranging from 0-6. A higher score reflects a better outcome.
Time Frame: Mean at baseline and 16 weeks
Measure: Mean (Standard Deviation); unit: completed categories
Arm/Group | LFR rTMS | Sham Treatment
Number analyzed (Participants) | 13 | 17
completed categories
  0 weeks | 5.5 (0.707) | 6 (0)
  16 weeks | 6 (0) | 6 (0)

6. Secondary Outcome: Cognitive Reasoning as Assessed by the Number of Errors Made on the Wisconsin Card Sorting Test (WCST)
Description: The participant points to choice on the screen and the tester manipulates the mouse to make the response. The participant tells the tester if he or she wants to change the response and the tester clicks on the screen. The score is the number of errors, ranging from 0-128. A higher score reflects a poorer outcome.
Time Frame: Mean at baseline and 16 weeks
Measure: Mean (Standard Deviation); unit: errors
Arm/Group | LFR rTMS | Sham Treatment
Number analyzed (Participants) | 13 | 17
errors
  Baseline | 26 (24.042) | 11 (5.354)
  16 weeks | 10.5 (2.881) | 8.667 (1.633)

7. Secondary Outcome: Cognitive Reasoning as Assessed by the Number of Correct Trials on the Wisconsin Card Scoring Test (WCST)
Description: The participant points to choice on the screen and the tester manipulates the mouse to make the response. The participant tells the tester if he or she wants to change the response and the tester clicks on the screen. The score is the number of correct trials, ranging from 0-128. A higher score reflects a better outcome.
Time Frame: Mean at baseline and 16 weeks
Measure: Mean (Standard Deviation); unit: correct trials
Arm/Group | LFR rTMS | Sham Treatment
Number analyzed (Participants) | 13 | 17
correct trials
  Baseline | 74.5 (14.849) | 68.857 (9.703)
  16 weeks | 67 (4.05) | 69.667 (8.981)

8. Secondary Outcome: Evaluation of Brain Injury as Assessed by the Trailmaking Test B Score
Description: The Trailmaking B score is the number of seconds spent connecting numbered circles (1-13) to circles containing letters of the alphabet (A-L) in alternating sequential order. A maximum of 300 seconds is allowed. Score ranges from 0-300. Higher score reflects poorer outcome.
Time Frame: Mean at baseline and 16 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | LFR rTMS | Sham Treatment
Number analyzed (Participants) | 13 | 17
seconds
  Baseline | 68.411 (32.106) | 71.432 (42.1)
  16 weeks | 56.439 (16.723) | 68.015 (25.023)

9. Secondary Outcome: Immediate Recall as Assessed by Hopkins Verbal Learning Test (HVLT)
Description: The Hopkins Verbal Learning Test (HVLT) consists of a 12-item word list, composed of four words from each of the three semantic categories. The subject is instructed to listen carefully as the examiner reads the word list and attempt to memorize the words. The word list is then read to the subject at the approximate rate of one word every 2 seconds. This is done for three trials. The number of correctly-recalled words in each trial is recorded (maximum of 12). The score is a sum of all the correctly-recalled words from each trial, for a maximum score of 36.
Time Frame: Mean at baseline and 16 weeks
Measure: Mean (Standard Deviation); unit: sum of correctly-recalled words
Arm/Group | LFR rTMS | Sham Treatment
Number analyzed (Participants) | 13 | 17
sum of correctly-recalled words
  Baseline | 23.077 (5.722) | 25.938 (5.285)
  16 weeks | 23.538 (7.287) | 25.5 (5.279)

10. Secondary Outcome: Delayed Recall as Assessed by Hopkins Verbal Learning Test (HVLT)
Description: The HVLT consists of a 12-item word list, composed of four words from each of the three semantic categories. The subject is instructed to listen carefully as the examiner reads the word list and attempt to memorize the words. The word list is then read to the subject at the approximate rate of one word every 2 seconds. This is done for three trials. After the third learning trial, the patient is read 24 words and is asked to say "yes" after each word that appeared on the recall list (12 targets) and "no" after each word that did not (12 distractors). Half of the distractors are drawn from the same semantic categories as the targets (related distractors) and half are drawn from other categories (unrelated distractors). The number of correctly-recalled words in each trial is recorded (maximum of 12 per trial). The score is the sum of all the correctly-recalled words from each trial, for a maximum of 36. T-scores are reported (average T-score of 50 (ranges 40-60)
Time Frame: Mean at baseline and 16 weeks
Measure: Mean (Standard Deviation); unit: T-score of correctly-recalled words
Arm/Group | LFR rTMS | Sham Treatment
Number analyzed (Participants) | 13 | 17
T-score of correctly-recalled words
  Baseline | 44.364 (10.604) | 43.071 (9.635)
  16 weeks | 49.111 (12.956) | 47.692 (5.836)

11. Secondary Outcome: Delayed Recall as Assessed by Brief Visual Memory Test (BVMT)
Description: BVMT is used to evaluate visuospatial memory abilities in neuropsychological populations. A visual display of six simple figures arranged in a 2 × 3 matrix on an 8 × 11 booklet is shown to participants for three consecutive 10-second trials. After each trial, participants are to draw as many designs as accurately as they can and in the correct location after a 25-minute delay filled with other distractor tasks. Scoring of the delayed recall is based on the accuracy of the drawings and the location of the figures. For each figure, one point is awarded to each satisfactory domain resulting in a maximum of 12-points per trial for a total score range of 0-36, with higher scores indicating a better outcome.
Time Frame: Mean at baseline and 16 weeks
Measure: Mean (Standard Deviation); unit: accurately-drawn figures
Arm/Group | LFR rTMS | Sham Treatment
Number analyzed (Participants) | 13 | 17
accurately-drawn figures
  Baseline | 9.23 (2.713) | 9.688 (3.005)
  16 weeks | 8.308 (3.066) | 8.813 (2.509)

12. Secondary Outcome: Immediate Recall as Assessed by Brief Visual Memory Test (BVMT)
Description: BVMT is used to evaluate visuospatial memory abilities in neuropsychological populations. A visual display of six simple figures arranged in a 2 × 3 matrix on an 8 × 11 booklet is shown to participants for three consecutive 10-second trials. After each trial, participants are to draw as many designs as accurately as they can and in the correct location. Scoring of the immediate recall is based on the accuracy of the drawings and the location of the figures. For each figure, one point is awarded to each satisfactory domain resulting in a maximum of 12-points per trial, for a total score ranging from 0-36, with a higher score reflecting a better outcome.
Time Frame: Mean at baseline and 16 weeks
Measure: Mean (Standard Deviation); unit: accurately-drawn figures
Arm/Group | LFR rTMS | Sham Treatment
Number analyzed (Participants) | 13 | 17
accurately-drawn figures
  Baseline | 22.846 (9.547) | 24.313 (7.355)
  16 weeks | 23.231 (8.833) | 21.438 (6.593)

13. Secondary Outcome: Evaluation of Brain Injury as Assessed by the Trailmaking Test A Score
Description: Trailmaking A is a psychological test with a score that is the number of seconds spent in connecting 25 numbered circles in sequential order. Score ranges from 0-150. Higher score reflects poorer outcome.
Time Frame: Mean at baseline and 16 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | LFR rTMS | Sham Treatment
Number analyzed (Participants) | 13 | 17
seconds
  Baseline | 27.725 (8.285) | 31.434 (10.02)
  16 weeks | 23.133 (5.8) | 30.027 (12.642)

14. Secondary Outcome: Mean Generalized Anxiety Disorder (GAD) - 7 Questionnaire
Description: The GAD-7 questionnaire is used as a screening tool and severity measure for generalized anxiety disorder. The scale ranges from 0 - 21.
  0-4 = normal 5-9 = mild 10-14 = moderate >15 = severe
Time Frame: Baseline, 4, 8, 12, and 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LFR rTMS | Sham Treatment
Number analyzed (Participants) | 13 | 17
units on a scale
  Baseline | 12.636 (4.61) | 12.75 (5)
  4 weeks | 7.5 (6.375) | 7.824 (5.028)
  8 weeks | 6.917 (6.417) | 7.588 (5.874)
  12 weeks | 6.923 (5.423) | 7.688 (5.594)
  16 weeks | 7.538 (6.603) | 7.412 (5.853)

15. Secondary Outcome: Mean Trauma Severity as Assessed by the Davidson Trauma Scale (DTS)
Description: The DTS is a 17-item self-reported measure that assesses the 17 Diagnostic and Statistical Manual IV (DSM-IV) symptoms of post-traumatic stress disorder (PTSD).
  Items are rated on 5-point frequency (0 = "not at all" to 4 = "every day") and severity scales (0 = "not at all distressing" to 4 = "extremely distressing").
  The DTS yields a frequency score (ranging from 0 to 68), severity score (ranging from 0 to 68), and total score (ranging from 0 to 136). The severity score will be used to assess this outcome.
Time Frame: Baseline, 4, 8, 12, and 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LFR rTMS | Sham Treatment
Number analyzed (Participants) | 13 | 17
units on a scale
  Baseline | 34.154 (30.306) | 41.706 (40.769)
  4 weeks | 15 (20.01) | 24.063 (33.657)
  8 weeks | 11.462 (20.711) | 17.294 (32.711)
  12 weeks | 14.833 (22.938) | 27.125 (33.478)
  16 weeks | 16 (29.243) | 18.647 (32.581)

16. Secondary Outcome: Mean Level of Fatigue as Assessed by Patient Sleep Quality Index (PSQI)
Description: The PSQI score scale ranges from 0-21. 0 = very good sleep quality 21 = very bad sleep quality A total score of "5" or greater is indicative of poor sleep quality (reflecting a higher level of fatigue)
Time Frame: Baseline, 4, 8, 12, and 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LFR rTMS | Sham Treatment
Number analyzed (Participants) | 13 | 17
units on a scale
  Baseline | 13.846 (3.848) | 13.688 (3.591)
  4 weeks | 10.23 (4.585) | 10.647 (4.133)
  8 weeks | 9.846 (4.356) | 10.176 (2.877)
  12 weeks | 9.5 (4.758) | 10.235 (4.161)
  16 weeks | 9.154 (4.913) | 9.625 (3.793)

17. Secondary Outcome: Mean Level of Fatigue as Assessed by the Epworth Sleepiness Scale (ESS)
Description: The ESS is used to determine the level of daytime sleepiness. It is a questionnaire composed of 8 questions. The participant answers each question on a scale of 0 to 3 (0=no sleepiness, 1= mild sleepiness, 2= moderate sleepiness, 3= severe sleepiness). The total score is the sum of all responses for a maximum score of 24. A higher score reflects increased sleepiness.
Time Frame: Baseline, 4, 8, 12, and 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LFR rTMS | Sham Treatment
Number analyzed (Participants) | 13 | 17
units on a scale
  Baseline | 9.769 (4.746) | 9.412 (6.81)
  4 weeks | 5.846 (4.896) | 7.563 (4.381)
  8 weeks | 5.923 (3.883) | 6.063 (3.586)
  12 weeks | 6.667 (5.015) | 7 (4.536)
  16 weeks | 6.077 (4.609) | 6 (3.857)

18. Secondary Outcome: Mean Cognitive Function as Assessed by the Montreal Cognitive Assessment (MOCA)
Description: MOCA is designed to assess cognitive impairment and Alzheimer's Disease. It is composed of the following:
  Visuospatial and Executive Functioning: 5 points Animal Naming: 3 points Attention: 6 points Language: 3 points Abstraction: 2 points Delayed Recall (Short-term Memory): 5 points Orientation: 6 points Education Level: 1 point is added to the test-taker's score if he or she has 12 years or less of formal education.
  Score ranges 0-31, with ≥ 26 being normal cognitive function. The lower the score, the greater the level of cognitive impairment.
Time Frame: Mean at baseline and 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LFR rTMS | Sham Treatment
Number analyzed (Participants) | 13 | 17
units on a scale
  Baseline | 25.769 (2.619) | 26.5 (3.141)
  16 weeks | 26 (3.342) | 26.875 (3.442)

19. Secondary Outcome: Presence of Neuropsychiatric Symptoms as Assessed by Neurobehavioral Rating Scale (NBRS)
Description: The NBRS is a 28-item interview which includes a test of orientation and memory for recent events, questions regarding emotional state, post-concussional symptoms, focused attention, and concentration (performing serial sevens), explanation of proverbs, tasks of planning and mental flexibility, and delayed recall of three objects presented at the beginning of a session. Observations are also made regarding the patient's fatigability, visible signs of anxiety, disinhibition, agitation, hostility, difficulties in expressive and receptive communication, and disturbance of mood. The balance of the items are rated according to the patient's performance on brief tasks and quality of answers to interview questions. Each of the 28 items are scored on a scale of 0 (not severe) to 6 (extremely severe), for a maximum score of 168. A higher score reflects increased severity of neuropsychiatric symptoms.
Time Frame: Mean at baseline, 4, 8, 12, and 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LFR rTMS | Sham Treatment
Number analyzed (Participants) | 13 | 17
units on a scale
  Baseline | 51.23 (5.89) | 56.125 (10.683)
  4 weeks | 40.545 (10.709) | 40.727 (7.837)
  8 weeks | 44.222 (12.498) | 42.786 (13.116)
  12 weeks | 43.222 (10.072) | 39.273 (9.056)
  16 weeks | 39.154 (11.866) | 40.375 (10.513)

20. Secondary Outcome: Presence of Post-concussive Symptoms as Assessed by the Rivermead Post-Concussion Questionnaire (RPQ)
Description: Participants are asked to rate the severity of 16 different symptoms over the past 24 hours, on a severity scale from 0 to 4 (0 = not experienced, 1 = no more of a problem, 2 = mild problem, 3 = moderate problem, 4 = severe problem). The 16 symptoms include: headaches, dizziness, nausea and/or vomiting, hyperacusis, sleep disturbance, fatigue, being irritable, feeling depressed, feeling frustrated, forgetfulness, poor concentration, taking longer to think, blurred vision, light sensitivity, double vision, restlessness. Score ranges from 0 to 64, with a higher score reflecting increased severity of post-concussive symptoms.
Time Frame: Mean at baseline, 4, 8, 12, and 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LFR rTMS | Sham Treatment
Number analyzed (Participants) | 13 | 17
units on a scale
  Baseline | 26.769 (8.719) | 23.125 (14.184)
  4 weeks | 11.833 (8.747) | 11.765 (9.451)
  8 weeks | 14.154 (11.753) | 11 (8.075)
  12 weeks | 12.75 (12.009) | 11.857 (10.369)
  16 weeks | 10.538 (7.817) | 14.294 (14.886)

21. Secondary Outcome: Fatigue Severity as Assessed by the Fatigue Severity Scale (FSS)
Description: The FSS is a 9-item questionnaire which measures the severity of fatigue and how it interferes with certain activities. The items are scored on a 7-point scale with 1=strongly disagree and 7=strongly agree. The score ranges from 9 to a maximum of 63. A higher score reflects greater fatigue severity.
Time Frame: Mean at baseline, 4, 8, 12, and 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LFR rTMS | Sham Treatment
Number analyzed (Participants) | 13 | 17
units on a scale
  Baseline | 28.308 (15.124) | 41.176 (11.975)
  4 weeks | 28.385 (15.788) | 23.375 (15.362)
  8 weeks | 20.769 (13.116) | 29.938 (16.643)
  12 weeks | 23.25 (11.787) | 27.286 (18.168)
  16 weeks | 21.23 (13.02) | 29 (17.274)

22. Secondary Outcome: Aggressive Behavior as Assessed by the Modified Overt Aggression Scale (MOAS)
Description: MOAS measures four types of aggressive behavior as witnessed in the past week. Each section consists of five items, with the first section regarding verbal aggression, the second section focusing on aggression against property, the third section measuring autoaggression, and the fourth section concerning physical aggression. Participants are asked to check each item that is true over the last week. Items are allocated 0, 1, 2, 3 or 4 point(s), and then all points for each selected item are summed. The maximum total for each section is 10 if all items are selected. Total score ranges from 0-40 with a higher score indicating more aggressive behavior.
Time Frame: Mean at baseline, 4, 8, 12, and 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LFR rTMS | Sham Treatment
Number analyzed (Participants) | 13 | 17
units on a scale
  Baseline | 2.308 (2.136) | 3 (4.016)
  4 weeks | 1.308 (1.377) | 1.118 (2.759)
  8 weeks | 0.692 (.855) | 0.471 (1.068)
  12 weeks | 1.417 (2.429) | 1 (1.932)
  16 weeks | 1.308 (2.213) | 0.706 (1.312)

23. Secondary Outcome: Overall Satisfaction With Life as Assessed by the Satisfaction With Life (SWL) Questionnaire
Description: The SWL is a 7-point Likert-style response scale. The possible range of scores is 5-35, with a score of 20 representing a neutral point on the scale. Scores between 5-9 indicate the respondent is extremely dissatisfied with life, whereas scores between 31-35 indicate the respondent is extremely satisfied.
Time Frame: Mean at baseline, 4, 8, 12, and 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LFR rTMS | Sham Treatment
Number analyzed (Participants) | 13 | 17
units on a scale
  Baseline | 14.231 (7.132) | 10.625 (4.015)
  4 weeks | 21.538 (8.511) | 18.471 (8.769)
  8 weeks | 22.231 (8.207) | 17.647 (9.88)
  12 weeks | 22 (8.524) | 17 (8.809)
  16 weeks | 23.923 (6.898) | 18.647 (9.367)

24. Secondary Outcome: Presence of Social Connections as Assessed by the Social Ties Checklist (STC)
Description: The STC reflects the level of social contact. The score ranges from 0-10, with 0= excellent contact, 10=no contact. A higher score reflects poorer social contact.
Time Frame: Mean at baseline, 4, 8, 12, and 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LFR rTMS | Sham Treatment
Number analyzed (Participants) | 13 | 17
units on a scale
  Baseline | 3.154 (1.573) | 4.563 (2.065)
  4 weeks | 3.077 (1.706) | 3.765 (1.855)
  8 weeks | 2.769 (1.536) | 3.471 (1.7)
  12 weeks | 2.846 (1.573) | 3.688 (2.243)
  16 weeks | 2.846 (1.676) | 3.471 (2.065)

ADVERSE EVENTS:
Time Frame: Participants were assessed at follow-up visits at 4 weeks, 8 weeks, 12 weeks, and 16 weeks. Any Adverse Event up to 16 weeks is reported.
Arm/Group | LFR rTMS | Sham Treatment
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 6/17 | 7/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LFR rTMS (N=17) | Sham Treatment (N=17)
Headache (Nervous system disorders) | 5 (12) | 5 (12)
Depression (Psychiatric disorders) | 1 (4) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (3)
Dizziness (Nervous system disorders) | 1 (1) | 1 (2)
Blurred Vision (Nervous system disorders) | 1 (1) | 0 (0)
Tiredness (Nervous system disorders) | 1 (1) | 0 (0)
Discomfort (Nervous system disorders) | 1 (1) | 1 (1)
Puff Face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Face Twitching (Nervous system disorders) | 0 (0) | 1 (2)
Eye Twitching (Nervous system disorders) | 1 (1) | 0 (0)
Sleep Problem (Nervous system disorders) | 1 (1) | 1 (4)
Other (Blood and lymphatic system disorders) | 2 (8) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-10-28): https://cdn.clinicaltrials.gov/large-docs/21/NCT02367521/Prot_SAP_000.pdf